CLINICAL TRIAL: NCT05201456
Title: LithoVue Elite (LVE) Registry
Brief Title: LithoVue Elite Registry
Acronym: LVE
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0701
Record Dates: First submitted 2021-11-19; First posted 2022-01-21 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Kidney Stone; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Pressure Monitoring: Subjects in this cohort will undergo ureteroscopic procedure using LithoVue Elite pressure monitoring single use flexible scope, real-time pressure monitoring technology, which will provide surgeons with intraluminal pressure data in the kidneys and ureter.
  Interventions: Device: LithoVue Elite System
- Non-Pressure Monitoring: Subjects in this cohort will undergo ureteroscopic procedure using LithoVue Elite Non-pressure monitoring single use flexible scope.
  Interventions: Device: LithoVue Elite System

INTERVENTIONS:
Device: LithoVue Elite System — The LithoVue Elite System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes. It can also be used in conjunction with endoscopic accessories to perform various diagnostic and therapeutic procedures in the urinary tract.

SUMMARY:
To obtain postmarket safety and efficacy data on Boston Scientific LithoVue™ Elite System.

DETAILED DESCRIPTION:
LithoVue Elite Registry is a post-market, multi-center, open label, non-randomized, prospective study to document the safety and efficacy data on Boston Scientific LithoVue™ Elite System.

LithoVue Elite System, includes the StoneSmart™ Connect Console (reusable capital/workstation) and a single-use, disposable ureteroscope device.

The LithoVue Elite System is intended to be used to visualize organs, cavities and canals in the urinary tract (urethra, bladder, ureter, calyces and renal papillae) via transurethral or percutaneous access routes. It can also be used in conjunction with endoscopic accessories to perform various diagnostic and therapeutic procedures in the urinary tract.

This is a post-market registry study. Any subject who meets eligibility criteria, intends to undergo a diagnostic and/or therapeutic procedure utilizing the LithoVue Elite System, and is willing to provide written informed consent, will be approached and considered for enrollment in the study. Data from diagnostic/therapeutic ureteroscopy procedure and standard of care post-ureteroscopy follow-up visits will be collected. These standard of care follow-up visits are expected to be scheduled within 120 days of the ureteroscopic procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject intends to undergo diagnostic and/or therapeutic procedure in the urinary tract with Boston Scientific LithoVue Elite System
2. Subject is able to accurately detect and report pain
3. Subject is willing and able to complete subject questionnaire at specified time points
4. Subject is willing and able to return for all follow-up visits

Exclusion Criteria:

1. Subject meets any of the contraindications per LithoVue Elite System Instructions/Directions for Use (IFU/DFU)
2. Subject meets any of the contraindications per any accessory devices that will be used in the ureteroscopy procedure
3. Investigator deems subject not suitable for the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 250 subjects will be enrolled at approximately 11 sites globally
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of Serious Adverse Device Effects - Primary Safety Endpoint | Up to 120 days of follow up
  Primary safety end point is the occurrence of Serious Adverse Device Effects (SADE) related to the LithoVue Elite System including, but not limited to urinary tract perforation and ureteral avulsion
Technical Success using LithoVue Elite System - Primary Effectiveness Endpoint | Procedure
  Primary effectiveness endpoint is the technical success using LithoVue Elite System, defined as:
  * Scope allows access to intended urinary anatomy (including utilization of active deflection and guidewire or access sheath)
  * Scope allows diagnostic and therapeutic tools, as identified in product labelling, to be utilized at target area, if applicable
  * Scope provides sufficient imaging for target visualization, (stone, calyx, etc.)
  * Scope provides real-time urinary system pressure measurements at target sites, if applicable
  Tool used will be a yes or no question on the case report form

SECONDARY OUTCOMES:
Occurrence of Procedure-Related Adverse Events and/or Adverse Device Effects Related to the LithoVue Elite System - Secondary Safety Endpoint | Up to 120 days of follow up
  Secondary safety endpoint is the occurrence of Procedure-related adverse events and/or adverse device effects related to the LithoVue Elite System

OTHER OUTCOMES:
Stone Free Rate - Additional Endpoint | Up to 120 days of follow up
  Stone clearance assessed by stone free rates (SFR), if applicable, at the follow-up visit
Surgeon Satisfaction with use of Scope - Additional Endpoint | Procedure
  Surgeon satisfaction on the use of scope will be measured on a 1-5 Likert scale
Post-operative Pain (Brief Pain Inventory (BPI)) - Additional Endpoint | Discharge, 7 days post procedure and 30 days post procedure
  Pain intensity and pain interference score on a scale of 0 to 10 as measured on the BPI
Post-operative Infection - Additional Endpoint | Up to 30 days post procedure
  Post-operative infection within 30 days of the procedure
Post-operative Systemic Inflammatory Response Syndrome (SIRS) - Additional Endpoint | Up to 30 days post procedure
  In subjects hospitalized post-procedure for infection, the complication will be characterized using the clinical measurements of the Systemic Inflammatory Response Syndrome (SIRS) score, if available. Subjects with a score ≥2 points meet the SIRS criteria
Post-operative Quick Sepsis Related Organ Failure Assessment (qSOFA) - Additional Endpoint | Up to 30 days post procedure
  In subjects hospitalized post-procedure for infection, sepsis information based on Quick Sepsis Related Organ Failure Assessment (qSOFA) score will be collected, if available.
  Urinary sepsis will be defined as a qSOFA score ≥2 points

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, Principal Investigator — Vancouver General Hospital

IPD SHARING:
Plan to Share IPD: No